CLINICAL TRIAL: NCT01475591
Title: Individually Tailored Web-based Multimodal Pain Rehabilitation in Primary Health Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luleå Tekniska Universitet (Other)
Collaborators: Norrbottens County Council (Other Government)
Responsible Party: Principal Investigator, Peter Michaelson, Senior lecturer, Luleå Tekniska Universitet
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REHSAM_NLL_LTU
Record Dates: First submitted 2011-11-01; First posted 2011-11-21 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Musculoskeletal Pain
Keywords: persistent neuromusculoskeletal pain; neck; shoulder; back-area; risk; longlasting; pain syndrome
MeSH Terms: conditions — Musculoskeletal Pain; Somatoform Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Multimodal rehabilitation (No Intervention): The arm intervention is just multimodal rehabilitation.
  Interventions: Behavioral: Web-based multimodal rehabilitation based on cognitive based principles

INTERVENTIONS:
Behavioral: Web-based multimodal rehabilitation based on cognitive based principles — The patient will be randomized to either the interventions group (multimodal pain rehabilitation with an added web-based multimodal rehabilitation with CBT-influences) or a control group (multimodal pain rehabilitation).

SUMMARY:
The aim is to evaluate effects of early individually tailored web-based multimodal rehabilitation for persons with musculoskeletal neck/shoulder and back disorders in primary health care. The aim is also to study if this early web-based pain rehabilitation program is more cost-effective than only multimodal rehabilitation. Randomization will be done at each primary health care centre after screening to 1) Multimodal pain rehabilitation with web-based education and coaching support or 2) multimodal pain rehabilitation. The investigators suggest a clear rehabilitation chain where a web-based program is developed,evaluated and ready to implement if it shows positive effects on work-ability and/or is cost-effective. The research and implementation will be performed in a close cooperation with Luleå University of Technology.

ELIGIBILITY:
Inclusion Criteria:

* With persistent neuromusculoskeletal pain from the neck/shoulder/back-area and/or fibromyalgia and a screening
* > 90 on Lintons´ questionnaire, The Örebro Musculoskeletal Pain Questionnaire (Linton & Halldén., 1998; Hockings et.al., 2008)
* Fluent in Swedish language
* Working, or in disposition to at least 25%

Exclusion Criteria are persons with:

* Dementia
* Restricted cognitive functioning
* Comorbidity which might prevent treatment participation
* Identified abuse, retirement pension
* Ongoing causal treatment
* Pregnancy
* Patients lacking internet attached computers in their home

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2011-10; Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Work ability | 4 month

SECONDARY OUTCOMES:
Pain rating | 12 month
  Pain-rating is measured on a visual analog-scale
Self-efficacy in relation to workability | 12 month
  Self-efficacy in relation to work-ability is measured by a questionnarie
General health | 12 month
  General health is measured with SF-36 and EQ-5D.
Functional status | 12 month
  Functional status is measured with Pain disability index.

CONTACTS AND LOCATIONS:
Overall Officials: Gunvor Gard, Professor, Principal Investigator — Luleå University of Technology
Locations (1):
- Primary health care centers in Norrbotten county council, Luleå, Norrbotten County, Sweden

REFERENCES:
- [Derived] Calner T, Nordin C, Eriksson MK, Nyberg L, Gard G, Michaelson P. Effects of a self-guided, web-based activity programme for patients with persistent musculoskeletal pain in primary healthcare: A randomized controlled trial. Eur J Pain. 2017 Jul;21(6):1110-1120. doi: 10.1002/ejp.1012. Epub 2017 May 2. PMID 28464364
- [Derived] Nordin CA, Michaelson P, Gard G, Eriksson MK. Effects of the Web Behavior Change Program for Activity and Multimodal Pain Rehabilitation: Randomized Controlled Trial. J Med Internet Res. 2016 Oct 5;18(10):e265. doi: 10.2196/jmir.5634. PMID 27707686